CLINICAL TRIAL: NCT07340346
Title: Evaluation of the Reliability of Preoperative Airway Assessment Tests in Predicting Difficult Airway Management in Obstetric Patients Undergoing Cesarean Section
Brief Title: Prediction of Difficult Airway in Cesarean Section Using Preoperative Airway Assessment Tests
Acronym: OB-DIFF-AIRWAY
Status: Completed | Type: Observational
Sponsor: Akdeniz University Hospital (Other)
Responsible Party: Principal Investigator, ALİ DEMİRTAŞ, Faculty Member, Department of Anesthesiology and Reanimation, Akdeniz University Hospital
Other Study IDs: Difficult Airway in Cesarean
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Difficult Airway; Airway Management; Obstetric Anesthesia
Keywords: Preoperative Airway Assessment; Mallampati Score; Difficult Intubation; Obstetric Patients
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstetric Patients Undergoing Cesarean Section: Adult obstetric patients undergoing elective or urgent cesarean section who received standard preoperative airway assessment as part of routine anesthetic care. Airway management was performed according to institutional clinical practice without any study-related intervention.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study. No experimental intervention was assigned. All assessments and airway management procedures were performed as part of routine clinical practice.

SUMMARY:
This observational study (OB-DIFF-AIRWAY: Obstetric Difficult Airway Study) aimed to evaluate the accuracy of commonly used preoperative airway assessment tests in predicting difficult airway management in obstetric patients undergoing cesarean section. Difficult airway remained a significant cause of anesthesia-related complications, particularly in pregnant patients due to physiological and anatomical changes.

Adult pregnant women scheduled for elective or urgent cesarean section underwent standard preoperative airway assessment, including Mallampati classification, thyromental distance, interincisor distance, neck circumference, and other routine clinical evaluations. Airway management during anesthesia was performed according to standard clinical practice. No additional intervention was applied for the purpose of the study.

The relationship between preoperative airway assessment findings and actual airway management difficulty was analyzed. The results of this study may help improve preoperative airway evaluation strategies and enhance patient safety in obstetric anesthesia.

DETAILED DESCRIPTION:
Difficult airway management is one of the most critical challenges in anesthetic practice and is associated with increased morbidity and mortality. Obstetric patients represent a particularly high-risk population due to pregnancy-related physiological changes such as airway edema, weight gain, reduced functional residual capacity, and increased oxygen consumption. Despite routine use of various preoperative airway assessment tests, their predictive value in obstetric patients remains controversial.

This prospective observational study was conducted to evaluate the reliability of commonly used preoperative airway assessment tests in predicting difficult airway management in patients undergoing cesarean section. The study was performed at Akdeniz University Hospital between August 23, 2023, and August 23, 2024.

Adult obstetric patients scheduled for elective or urgent cesarean section under anesthesia were included. Patients with known airway pathology, prior difficult airway history requiring advanced airway techniques, or incomplete airway assessment data were excluded according to predefined criteria.

Preoperative airway assessment was performed as part of routine anesthetic evaluation and included Mallampati classification, thyromental distance, interincisor distance, neck circumference, and other standard clinical parameters. No additional procedures or interventions were introduced for research purposes. Anesthetic management and airway techniques were determined by the attending anesthesiologist in accordance with institutional standards.

Airway management difficulty was recorded intraoperatively based on predefined clinical criteria, including difficulty with mask ventilation, laryngoscopy, or tracheal intubation. The association between preoperative airway assessment findings and observed airway difficulty was analyzed using appropriate statistical methods. Difficult airway management was defined as the presence of at least one of the following predefined intraoperative criteria:

difficult mask ventilation (Han classification ≥ 3), difficult laryngoscopy (Cormack-Lehane grade III-IV), or failure of tracheal intubation on the first attempt.

Patients were enrolled using a consecutive non-probability sampling approach, including all eligible obstetric patients undergoing cesarean delivery during the study period.

The sample size was determined by the consecutive inclusion of all eligible patients undergoing cesarean delivery at the study center during the predefined study period.

The primary objective of the study was to assess the predictive value of individual and combined airway assessment tests for difficult airway management in obstetric patients. Secondary objectives included identifying potential risk factors associated with airway difficulty and evaluating the overall incidence of difficult airway in the study population.

The findings of this study are expected to contribute to improved preoperative airway evaluation and risk stratification in obstetric anesthesia, thereby enhancing patient safety and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult obstetric patients aged 18 years or older
* Scheduled for elective or urgent cesarean section
* Undergoing routine preoperative airway assessment
* Provided written informed consent

Exclusion Criteria:

* Known congenital or acquired airway pathology
* History of difficult airway requiring advanced airway techniques
* Emergency situations requiring immediate airway management without standard preoperative assessment
* Incomplete or missing airway assessment data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult pregnant women aged 18 years and older who underwent elective or urgent cesarean section at a tertiary university hospital. All participants received standard preoperative airway assessment as part of routine anesthetic care.
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Prediction of Difficult Airway Using Preoperative Airway Assessment Tests | During anesthesia induction
  The primary outcome is the ability of preoperative airway assessment tests to predict difficult airway management during cesarean delivery.
  Predictive performance was evaluated using sensitivity, specificity, positive and negative predictive values, and the area under the receiver operating characteristic (ROC) curve (AUC).
  Difficult airway was defined based on predefined intraoperative criteria such as difficulty in mask ventilation, difficult laryngoscopy, or difficult tracheal intubation as assessed by the attending anesthesiologist.

SECONDARY OUTCOMES:
Incidence of Difficult Airway in Obstetric Patients | During anesthesia induction
  The incidence of difficult airway management among obstetric patients undergoing cesarean section was evaluated based on predefined clinical criteria.
Association Between Individual Airway Assessment Tests and Difficult Airway | During anesthesia induction
  The association between individual preoperative airway assessment tests and the occurrence of difficult airway management was analyzed to identify potential risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: ALİ DEMİRTAŞ, Principal Investigator — Akdeniz University Hospital
Locations (1):
- Akdeniz University Hospital, Antalya, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mushambi MC, Jaladi S. Airway management and training in obstetric anaesthesia. Curr Opin Anaesthesiol. 2016 Jun;29(3):261-7. doi: 10.1097/ACO.0000000000000309. PMID 26844863
- [Background] Freedman RL, Lucas DN. MBRRACE-UK: saving lives, improving mothers' care - implications for anaesthetists. Int J Obstet Anesth. 2015 May;24(2):161-73. doi: 10.1016/j.ijoa.2015.03.004. Epub 2015 Mar 14. PMID 25841640
- [Background] McKeen DM, George RB, O'Connell CM, Allen VM, Yazer M, Wilson M, Phu TC. Difficult and failed intubation: Incident rates and maternal, obstetrical, and anesthetic predictors. Can J Anaesth. 2011 Jun;58(6):514-24. doi: 10.1007/s12630-011-9491-9. Epub 2011 Apr 7. PMID 21472485